CLINICAL TRIAL: NCT06158802
Title: Evaluation of Human Papillomavirus Vaccine Coverage in Girls and Young Women With Chronic Disease
Acronym: MC-HPV
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210417; 2021-A02421-40 (Other: IDRCB number)
Record Dates: First submitted 2023-11-24; First posted 2023-12-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Human Papillomavirus Vaccine; Chronic Condition
Keywords: Human papillomavirus vaccine; Young women with chronic condition; Vaccination coverage rate
MeSH Terms: conditions — Chronic Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic condition: Girls and young women between the ages of 11 and 20 suffering from chronic condition
  Interventions: Other: Questionnaire
- Control: Girls and young women between the ages of 11 and 20 in good health
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire on human papillomavirus vaccine status of girls and young women and modalities of the vaccination or reason of the non-vaccination.
  The questionnaire is completed by the patient.

SUMMARY:
The main objective of the study is to determine the vaccination coverage rate for human papillomavirus in adolescents aged 11 to 20 with chronic disease and treated at the Necker-Enfants Malades Hospital, compared to a population witnessed adolescent girls aged 11 to 20 years without chronic disease.

DETAILED DESCRIPTION:
Girls and young women with chronic condition are at higher risk for infections that can be prevented by vaccination. Human papillomavirus infection is very common, one of the three most common in the general population. A vaccine exists to significantly prevent this infection and its complications.

In France, it is advisable to vaccinate girls and boys from the age of 9 years and as soon as possible in the case of acquired immunodeficiency since these patients are more likely to be suffering from cancer induced by the human papillomavirus.

In France, the overall rate of vaccination coverage for girls is 21%, which is significantly lower than in several other industrialized countries.

The vaccination coverage rate for human papillomavirus in patients with chronic diseases may be even lower.

The main objective of the study is to determine the vaccination coverage rate for human papillomavirus in adolescents aged 11 to 20 with chronic condition and treated at the Necker-Enfants Malades Hospital, compared to a population witnessed adolescent girls aged 11 to 20 years without chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* Information and non-opposition of major patients and holders of parental authority of minor patients and minor patients
* Girls and young women aged 11 to 20
* To be followed at the Necker-Enfants Malades Hospital ("chronic condition" group)
* To be followed at the Specialized Medical Center for Children and Adolescents ("control" group)
* Have a chronic condition ("chronic condition" group) :

  * Diabetes type 1
  * Metabolic diseases
  * Patients followed in immuno-hematology
  * Cystic Fibrosis
  * Sickle
  * Kidney transplant
  * Heart Disease
  * Inflammatory bowel diseases
  * Rare anorectal and pelvic anomalies
* Live in France
* Comprehension of the French language (oral and written)

Exclusion Criteria:

* Have a contraindication to the HPV vaccine - Gardasil 9 (Vidal Hoptimal, 2018)
* Have a contraindication to the HPV vaccine - Gardasil (Vidal Hopitmal, 2018)
* Have a contraindication to HPV vaccine - Cervarix (Vidal Hoptimal, 2018)

Ages: 11 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Patients aged from 11 to 20 to cover the recommended age window for HPV vaccination, ie between 11 and 14 years old, with the possibility of catching up between 15 and 19 years of age (Public Health France, 2019).
  "Chronic condition" group: type 1 diabetes, metabolic diseases, immuno-hematological diseases, cystic fibrosis, sickle cell disease, kidney transplant, heart disease and inflammatory bowel disease, rare anorectal and pelvic malformations. Recruitment at the Necker-Enfants Malades Hospital and at the Specialized Medical Center for Children and Adolescents in Paris.
  "Control" group: patients in good health. Recruitment at the Specialized Medical Center for Children and Adolescents in Paris.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Immunization coverage rate for human papillomavirus vaccine | Day 1
  Percentage of patients with or without a chronic illness who have received HPV vaccination (complete vaccination schedule).

SECONDARY OUTCOMES:
Intention of vaccination by human papillomavirus vaccine by the usual health professionals | Day 1
  Percentage of patients with or without a chronic illness who have been offered HPV vaccination.
Category of health professionals offering vaccination by human papillomavirus vaccine | Day 1
  Patients with or without a chronic illness to whom vaccination has been offered/prescribed :
  * Percentage of vaccination offered/prescribed by the general practitioner
  * Vaccination percentage proposed/prescribed by the pediatrician,
  * Vaccination percentage proposed/prescribed by the gynecologist,
  * Percentage of vaccination proposed/prescribed by the specialist doctor,
  * Percentage of vaccination offered/prescribed by another healthcare professional.
Reasons for non-vaccination by human papillomavirus vaccine | Day 1
  Patients suffering from a chronic illness or not and not vaccinated:
  * Percentage of patients not vaccinated due to fear/apprehension,
  * Percentage of patients not vaccinated because they did not know this vaccine,
  * Percentage of patients not vaccinated because they are against vaccination,
  * Percentage of patients not vaccinated due to lack of time.
Description of parameters that may impact vaccination coverage for human papillomavirus vaccine | Day 1
  Description of patients with or without a chronic illness and vaccinated or not against HPV
  * Average age of patients at the time of inclusion,
  * Socio-professional category of parents (father's and mother's profession),
  * Average age at menarche,
  * Assessment of risk behaviors (percentage of patients who smoke, percentage of patients who consume alcohol),
  * Percentage of patients who have started their sexual life,
  * Average age at first sexual intercourse,
  * Percentage of patients followed by a pediatrician,
  * Percentage of patients followed by a general practitioner,
  * Percentage of patients followed by a gynecologist.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina DA COSTA, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Alaa CHEIKHELARD, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Centre Médical Spécialisé de l'Enfant et de l'Adolescent (CMSEA), Paris
  - Hôpital Necker-Enfants Malades, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofstetter AM, Camargo S, Natarajan K, Rosenthal SL, Stockwell MS. Vaccination Coverage of Adolescents With Chronic Medical Conditions. Am J Prev Med. 2017 Nov;53(5):680-688. doi: 10.1016/j.amepre.2017.07.017. Epub 2017 Sep 18. PMID 28928039
- [Background] Gras-Le Guen C, Legrand A, Caquard M, Micaelli X, Picherot G, Lacroix S, Volteau C, Launay E. Chronically ill adolescents are also incompletely vaccinated: A cross-sectional study in France. Vaccine. 2017 Aug 24;35(36):4707-4712. doi: 10.1016/j.vaccine.2017.07.042. Epub 2017 Jul 29. PMID 28760611
- [Background] Hoffman L, Okcu MF, Dreyer ZE, Suzawa H, Bryant R, Middleman AB. Human papillomavirus vaccination in female pediatric cancer survivors. J Pediatr Adolesc Gynecol. 2012 Oct;25(5):305-7. doi: 10.1016/j.jpag.2012.05.004. Epub 2012 Jul 24. PMID 22831900